CLINICAL TRIAL: NCT02071602
Title: CD-NP (Cenderitide) Therapy for the Preservation of Left Ventricular Function Post Anterior Myocardial Infarction - Pilot Study
Brief Title: CD-NP (Cenderitide) Therapy for the Preservation of Left Ventricular Function
Acronym: BELIEVE III
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Horng Chen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-006317
Record Dates: First submitted 2013-11-15; First posted 2014-02-26 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction of Anterior Wall
Keywords: Heart attack; Myocardial Infarction; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — cenderitide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo infused for up to 72 hours IV
  Interventions: Drug: CD-NP
- CD-NP 5 ng/kg/min (Active Comparator): CD-NP 5 ng/kg/min infused for up to 72 hours IV
  Interventions: Drug: CD-NP
- CD-NP 10 ng/kg/min (Placebo Comparator): CD-NP 10 ng/kg/min infused for up to 72 hours IV
  Interventions: Drug: CD-NP

INTERVENTIONS:
Drug: CD-NP — Randomized 1:1:1
  Other Names: Cenderitide

SUMMARY:
The primary endpoint is to assess the safety and tolerability of Cenderitide (CD-NP) with the incidence of symptomatic hypotension being one of the key safety variables.

DETAILED DESCRIPTION:
This is a "proof of concept", randomized, double-blind, placebo controlled study. The study population will include 60 patients admitted with a first time ST elevation anterior STEMI as diagnosed by the following criteria: a) Significant chest discomfort and /or shortness of breath; b) ST segment elevation (1.5 mV total) in two or more adjacent anterior precordial leads; c) Successful reperfusion therapy (>TIMI grade 2 flow) either with thrombolytics or PTCA within 24 hours of onset of symptoms as documented by coronary angiography; and d) No previous history of an anterior AMI or previous ECG suggesting an old anterior AMI.

Patients will be randomized to one of two doses of CD-NP (5 ng/kg/min and 10 ng/kg/min) or placebo continuous infusion for up to 72 hours in a 1:1:1 manner. All patients will receive other standard medical therapies as determined appropriate by the physician and in accordance to the ACC/AHA guidelines

ELIGIBILITY:
Inclusion Criteria:

* Significant chest discomfort and /or shortness of breath
* ST segment elevation (1.5 mV total) in two or more adjacent anterior precordial leads
* Successful reperfusion therapy (>TIMI grade 2 flow) either with thrombolytics or any mechanical forms of revascularization, including stent, PTCA, thrombectomy, etc. within 24 hours of onset of symptoms as documented by coronary angiography
* No previously known history of AMI (prior to current cardiac event) or no previous ECG (prior to current cardiac event) suggesting an old AMI (Q wave on presenting ECG is not an exclusion)..

Exclusion Criteria:(Assessed at the time of enrollment unless otherwise stated)

* Cardiogenic shock, acute heart failure or hypotension (Systolic BP < 90 mmHg)
* Previous known decreased EF < 40%
* Atrial Fibrillation
* Persistent signs and symptoms of Post MI ischemia
* Requirement of pressors for maintenance of blood pressure.
* Intra-aortic blood pump use
* Significant (moderate-severe) valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension.
* Severe congenital heart diseases
* Sustained ventricular tachycardia or ventricular fibrillation
* Second or third degree heart block without a permanent cardiac pacemaker
* Stroke within 3 months or other evidence of significantly compromised CNS perfusion
* Total bilirubin of > 2.5 mg/dL or other liver enzymes >2.5 times the upper limit of normal if available clinically and measured within the last 7 days
* Patients with calculated GFR <30 ml by MDRD equation or those with acute kidney injury as defined by an increase of plasma creatinine of 0.5 mg/dL from a plasma creatinine measured within the last 7 days
* Serum sodium of < 125 mEq/dL or > 160 mEq/dL if available clinically and measured within the last 7 days
* Serum potassium of < 3.0 mEq/dL or > 5.8 mEq/dL if available clinically and measured within the last 7 days
* Hemoglobin < 8.5 gm/dl if available clinically and measured within the last 7 days
* Other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data
* Received an investigational drug within 1 month prior to dosing
* Female subject who is pregnant or breastfeeding
* In the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2018-05 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with symptomatic hypotension | baseline to 30 days

SECONDARY OUTCOMES:
Comparison of LV function improvement between placebo vs. CD-NP groups | baseline to 30 days
Exploratory analyses of Major Adverse Cardiovascular Events (MACE) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Horng Chen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Related Info — https://www.mayo.edu/research/clinical-trials